CLINICAL TRIAL: NCT01048528
Title: Phase II Study of Stress Management and Vaccine Response Among Women at Risk for Breast Cancer
Brief Title: Health SMART (Stress Management and Relaxation Training)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Bonnie A. McGregor, PhD / Assistant Member, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-6940; 1R21CA134813 (NIH)
Record Dates: First submitted 2009-11-03; First posted 2010-01-13 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: immune response to vaccines; stress management; perceived risk for breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress Management (Experimental): Stress Management and Relaxation Training workshops
  Interventions: Behavioral: Cognitive Behavioral Stress Management (CBSM)
- Wait-list (No Intervention): Wait-list comparison group

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management (CBSM) — The intervention employs CBSM techniques interwoven with information in a supportive group format. The information portion of the intervention focuses on learning to cope with daily stressors, and learning about optimal use of social support. Avoidance coping is discouraged, and acceptance and reframing are instead encouraged as coping responses. Health behavior change, framed as a coping technique, will also be discussed using motivational interviewing techniques. Relaxation techniques include progressive muscle relaxation, guided imagery, autogenics, meditation, and deep breathing. The goal of the CBSM intervention is thus to reduce distress through a variety of techniques.
  Other Names: Stress Management and Relaxation Training (SMART)
  Arms: Stress Management

SUMMARY:
The study will examine the effects of a cognitive behavioral stress management (CBSM) group intervention on antibody and cellular immune function among women who are at elevated risk for breast cancer because of family history.

Hypothesis 1: Women who participate in the CBSM intervention will have a larger primary and secondary antibody response to HA vaccine compared to women in the comparison group.

Hypothesis 2: In response to stimulation with HA antigen, lymphocytes from women who participate in the CBSM intervention will have larger primary and secondary in-vitro proliferative response to HA antigen, and increased primary and secondary in-vitro TH1 cytokine response to HA antigen compared to lymphocytes from women in the comparison group.

Hypothesis 3: Women who participate in the 10-week CBSM group intervention will report lower levels of distress immediately after the intervention compared to women in the comparison group. Changes in distress as a result of the intervention will be associated with any significant changes in immune function discovered in Aims 1 and 2.

DETAILED DESCRIPTION:
Cancer vaccines are emerging as important tools for cancer treatment and prevention. Unfortunately, the cohorts that ultimately will benefit most from the vaccines, those at elevated risk for cancer, are likely to be stressed. Chronic stress can impair immune function, including immune response to vaccines. An inadequate response to vaccines can weaken their protective effect. Women at elevated risk for breast cancer can experience significant levels of distress and have associated immune function decrements. Interventions to treat distress-related immune decrements among these women are needed because these women will be among the first candidates for breast cancer vaccines. In theory, stress-management interventions should improve immune function and response to vaccines; however, the findings to date are mixed. The proposed investigation will conduct an exploratory randomized clinical trial to collect preliminary data on the efficacy of a cognitive behavioral stress management (CBSM) group intervention among women who are at elevated risk for breast cancer because of family history and who are reporting elevated levels of distress. Study outcomes will include antibody and cellular immune response to hepatitis A vaccine and self-reported distress.

ELIGIBILITY:
Inclusion Criteria:

* Family history of breast cancer
* Fluent in English
* Working phone and address
* Plan to live in the area for one year
* Reporting elevated levels of distress at screening.

Exclusion Criteria:

* Prior cancer diagnosis (except non-melanoma skin cancer)
* Current major depressive episode
* History of Bipolar Disorder or Schizophrenia
* History of autoimmune disease
* History of Hepatitis A or HA vaccination
* Use of immune modulating drugs (e.g. corticosteroids, antihistamines), nicotine, or > 3 drinks/ day alcohol

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Linear mixed models regression with an exchangeable covariance structure will be used to determine the average change in IgM, IgG and proliferative response to HA vaccine antibody response to HA vaccine following the intervention, as a function of time. | From post-intervention to 1-month post-intervention (primary antibody response) and from 6-months post-intervention to 7-months post-intervention (secondary antibody response)

SECONDARY OUTCOMES:
Linear mixed model regression with an exchangeable covariance structure will be used to investigate the effects of change in distress on immune response as a function of time. We will include time as a random effect. | Length of the protocol (Basline to 7 months post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie A. McGregor, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Sannes TS, Dolan E, Albano D, Ceballos RM, McGregor BA. Stress management reduces intraindividual cortisol variability, while not impacting other measures of cortisol rhythm, in a group of women at risk for breast cancer. J Psychosom Res. 2015 Nov;79(5):412-9. doi: 10.1016/j.jpsychores.2015.09.012. Epub 2015 Sep 28. PMID 26526317